CLINICAL TRIAL: NCT04192721
Title: Controlled, Randomized, Cognitive Behavioral Therapy-Based Group Counseling for Nursing Students With Depressive Symptoms
Brief Title: Cognitive Behavioral Therapy-Based Group Counseling
Acronym: CBTBGC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Satı Demir, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDemir
Record Dates: First submitted 2019-11-28; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Depression Moderate; Depression Mild
Keywords: depression; cognitive behavioral therapy; group counseling; nursing students
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The study used a randomized control clinical trial design. In the BDI pre-test, 80 of the students with mild or moderate depressive symptoms met the other inclusion criteria of the study and volunteered to participate in the study. Out of 80 participants, 40 were randomly assigned to the intervention group and 40 to the control group using computer-generated random number sequences. The study was completed with a total of 63 participants (n=31 for the intervention group; n=32 for the control group). While CBT-based group counseling was given to the intervention group, no counseling was given to the control group during the study.
  The participants were evaluated at three time points: at screening (pre-test), six weeks after screening (post-intervention/post-test), and two months after the post-test. The measurements were taken simultaneously in the intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy-Based Group Counseling (Experimental): The CBT-based group counseling provided to the intervention group was carried out as a group intervention with structured sessions in which various techniques and methods of CBT, having mainly educational content, were applied, including an experiential interaction process. The counseling was performed in a total of six 60- to 90-minute sessions, comprising one session per week for four groups consisting of six to 10 members each.
  Interventions: Behavioral: Cognitive Behavioral Therapy-Based Group Counseling
- Control group (No Intervention): No counseling was given to the control group during the study.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy-Based Group Counseling — * Relaxation techniques
  * Providing personal development books
  * Sharing the factors affecting the situation defined as depression (brainstorming)
  * Explaining the link between depressive symptoms, thoughts, feelings, and behaviors
  * Explaining automatic thoughts
  * Application of relaxation techniques; deep-breathing exercises
  * Identifying alternative thoughts
  * Explaining the correlation between alternative thoughts and mood
  * Introduction of the Automatic-Thought Registration Form and distribution to students
  * Describing the effects of depression on social interaction
  * Explaining activities that could be done individually and with the group
  * Distribution of the activity list to students
  * Description of ways of coping with stress
  * Determination of individual stressors and their effects
  * Planning for the future: preventing depression
  * Discussion of assumptions/expectations about life
  * Homeworks related to session contents
  Arms: Cognitive Behavioral Therapy-Based Group Counseling

SUMMARY:
The university environment presents a valuable opportunity to reach the young population of society, which has a high risk of depression, and to provide protective mental-health services. This study aimed to evaluate the effectiveness of cognitive behavioral therapy-based group counseling focused on the depressive symptoms, anxiety levels, automatic thoughts, and coping ways among undergraduate nursing students with mild to moderate depressive symptoms.

DETAILED DESCRIPTION:
This study aimed to evaluate the effectiveness of cognitive behavioral therapy-based group counseling focused on the depressive symptoms, anxiety levels, automatic thoughts, and coping ways among undergraduate nursing students with mild to moderate depressive symptoms.

The study was completed with a total of 63 participants (n=31 for the intervention group and n=32 for the control group) in the 2017-2018 academic year. The effect of the intervention was evaluated with the Beck Depression Inventory, Beck Anxiety Inventory, Automatic Thoughts Questionnaire, and Ways of Coping Questionnaire. The measurements were taken 3 times: pre-test, post-test, and 2-months post-test.

ELIGIBILITY:
Inclusion Criteria:

* Having mild depressive symptoms according to the BDI
* Having moderate depressive symptoms according to the BDI
* Being native speakers of Turkish
* Agreeing to participate in the entire intervention process

Exclusion Criteria:

* Having substance abuse
* Having another psychiatric diagnosis
* Using psychotropic drugs
* Receiving other counseling or therapy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) | Change from baseline to 6 weeks (also assessed at 14 weeks post-baseline)
  It measures the risk level of depression. It has 21 items. Each item is scored 0-3 points and the total score ranges from 0-63 (0-9=no; 10-16= mild; 17-20= moderate; 21-26=high; 27 or more points severe depressive symptoms)
Beck Anxiety Inventory (BAI) | Change from baseline to 6 weeks (also assessed at 14 weeks post-baseline)
  This self-assessment scale determines anxiety level. It consists of 21 items. Each item is scored 0-3 points and the total score ranges from 0-63. As the total score increases, the anxiety level increases.
Automatic Thoughts Questionnaire (ATQ) | Change from baseline to 6 weeks (also assessed at 14 weeks post-baseline)
  It measures the thought patterns and negative self-assessments commonly seen in depression. It consists of 30 items. Each item is scored 1-5 points and the total score ranges from 30-150 points. A high score indicates that the frequency of automatic thoughts related to depression is high.
Ways of Coping Questionnaire (WCQ) | Change from baseline to 6 weeks (also assessed at 14 weeks post-baseline)
  It measures the thought patterns and negative self-assessments commonly seen in depression. It consists of 30 items. Each item is scored 1-5 points and the total score ranges from 30-150 points. A high score indicates that the frequency of automatic thoughts related to depression is high.

CONTACTS AND LOCATIONS:
Overall Officials: Satı Demir, PhD, Principal Investigator — Gazi University Health Sciences Faculty, Ankara, Turkey
Locations (1):
- Satı Demir, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Other researchers will be able to read detailed information such as the research method and results when the research is published. The "Research Protocol" will be available on the this PRS page.